CLINICAL TRIAL: NCT03312842
Title: A Phase Ia/Ib, Open-Label, Multiple-Dose, Dose-Escalation and Expansion Study of the Anti-PD-L1 Monoclonal Antibody CS1001 in Subjects With Advanced Solid Tumors
Brief Title: A Phase Ia/Ib Study of CS1001 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1001-101
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CS1001 (Experimental)
  Interventions: Drug: CS1001

INTERVENTIONS:
Drug: CS1001 — In the dose escalation part, the dose levels will be escalated following a modified 3+3 dose escalation scheme.
  In the dose expansion part, patients will be assigned to different groups based on their tumor type.

SUMMARY:
This is a phase Ia/Ib, open-label, multiple-dose, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of CS1001 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. With advanced-stage or metastatic tumor (unresectable) and experienced progression since last anti-tumor treatment; standard therapy is not available or rejected.
2. ECOG performance status of 0 or 1.
3. Subjects must have at least one measurable lesion.
4. Patients with life expectancy ≥ 3 months.
5. Subject must have adequate organ function.
6. Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for six months after last study drug administration.

Exclusion Criteria:

1. Known brain metastasis or other CNS metastasis that is either symptomatic or untreated.
2. Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded.
3. Patients who have received immune checkpoint proteins/antibody/medicine (including PD-1, PD-L1, etc) for treatment.
4. Known history of HIV infection.
5. Hepatitis B surface antigen (HBsAg) and Hepatitis B core antibody (HBcAb) positive or Hepatitis C virus (HCV) antibody positive.
6. Patients who have serious hypersensitive reaction to monoclonal antibodies, and have history of uncontrolled allergic asthma.
7. Known history of alcoholism or drugs abuse.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CS1001 | From first dose to 30 days after last dose of CS1001, up to 2 years
To determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of CS1001 | From first dose to 30 days after last dose of CS1001, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Gong J, Cao J, Zhang Q, Xu N, Zhao Y, Xing B, Miao Z, Wu Y, Pan H, Gao Q, Li X, Liu B, Li W, Pei Z, Xia H, Qi Q, Dai H, Shi Q, Yang J, Li J, Shen L. Safety, antitumor activity and biomarkers of sugemalimab in Chinese patients with advanced solid tumors or lymphomas: results from the first-in-human phase 1 trial. Cancer Immunol Immunother. 2022 Aug;71(8):1897-1908. doi: 10.1007/s00262-021-03102-3. Epub 2022 Jan 5. PMID 34984540